CLINICAL TRIAL: NCT04750460
Title: The Effect of Teriparatide on the Early Postoperative Hypocalcemia After Parathyroidectomy in Dialysis Patients: a Pilot, Randomized Trial
Brief Title: Injection of Teriparatide to Prevent Hypocalcemia After Parathyroidectomy in Dialysis Patients (TeriCa).
Acronym: TeriCa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Novokshonov Konstantin, MD, PHD, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TeriCa
Record Dates: First submitted 2021-02-02; First posted 2021-02-11 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease-Mineral and Bone Disorder; Dialysis; Hypocalcemia; Hypoparathyroidism
Keywords: Parathyroidectomy; Teriparatide; Parathyroid hormone
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Chronic Kidney Disease-Mineral and Bone Disorder; Hypocalcemia; Hypoparathyroidism | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teriparatide group (11 patients) (Experimental): Dialysis-dependent patients underwent total parathyroidectomy with autotransplantation of parathyroid tissue, who will receive subcutaneous injections ot recombinant parathyroid hormone (Teriparatide) after surgery in addition to the standard local protocol for hypocalcemia treatment.
  Interventions: Drug: Teriparatide
- Control group (9 patients) (No Intervention): Dialysis-dependent patients underwent total parathyroidectomy with autotransplantation of parathyroid tissue, receiving standard local protocol for hypocalcemia treatment (2 micrograms of alphacalcidol plus 4 grams of oral calcium daily).

INTERVENTIONS:
Drug: Teriparatide — Subcutaneous injections of study drug will be assigned immediately after parathyroidectomy (20 mcg), on the 1st (20 mcg) and 2nd (10 mcg) postoperative day.
  Other Names: Forsteo
  Arms: Teriparatide group (11 patients)

SUMMARY:
This is a pilot randomized controlled trial aimed to evaluate the effect of teriparatide on the clinical course of hypocalcemia after parathyroidectomy for secondary hyperparathyroidism in dialysis-dependent patients.

DETAILED DESCRIPTION:
Postoperative hypocalcemia is a common complication after parathyroidectomy (PTx) for secondary hyperparathyroidism in dialysis-dependent patients. It is known to be associated with significant drop of parathyroid hormone (iPTH) level after surgery. Thus, in the present study we test the hypothesis that reducing iPTH difference before/after PTx with teriparatide injections immediately after surgery may alleviate clinical course of post-PTx hypocalcemia.

This is a feasible study aimed to determine the sample size for further large-scale trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years;
2. Patients with end-stage renal disease (ESRD) receiving hemodialysis or peritoneal dialysis treatment > 3 months prior surgery;
3. Severe secondary hyperparathyroidism defined as iPTH level > 800 pg/ml, followed with hypercalcemia and/or hyperphosphatemia; with presence of one or more nodular or diffuse parathyroid hyperplasia confirmed with CT;
4. Performed total parathyroidectomy with autotransplantation of the parathyroid tissue.

Exclusion Criteria:

1. Emergency surgery;
2. Primary hyperparathyroidism as a cause of ESRD;
3. Scheduled (before surgery) blood transfusion;
4. Re-operative surgery;
5. Known allergy to the study drug.
6. Malignant neoplasms of bone tissue (primary or metastatic).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Total serum calcium level | Day 1,2,3,4,5

SECONDARY OUTCOMES:
Parathyroid hormone level | Day 1, 2, 3, 4, 5
Serum phosphorus level | Day 1, 2, 3, 4, 5
Serum total alkaline phosphatase level | Day 1, 2, 3, 4, 5
Total serum calcium level | Day 2, 3, 4, 5
Ionized serum calcium level | Day 1, 2, 3, 4, 5
Serious adverse events (major cardiovascular events, fractures, arrhythmia episodes, death) | up to 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Petersburg State University Hospital, Saint Petersburg, Russia